CLINICAL TRIAL: NCT02358837
Title: Improving Breast Cancer Diagnostics by Novel Sonographic Techniques
Brief Title: Improving Breast Cancer Diagnostic by Novel sonographicTechniques Study
Acronym: RadioUS
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 204.08.2011
Record Dates: First submitted 2015-01-12; First posted 2015-02-09 (Estimated); Last update posted 2018-05-16 (Actual); Status verified 2018-05

CONDITIONS: Breast Cancer
Keywords: elastosonography; comparing conventional sonography with ductosonography
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Conventional Sonography: Conventional Sonography to detect breast lesion
- Ductosonography Technique: Ductosonography Technique to detect breast lesion

SUMMARY:
With the proposed project we seek to advance the detection and diagnosis of breast cancer in an outpatient breast clinic. Novel sonographic approaches will be scrutinized. The first aim of this study will be to explore whether there is an advantage of ductosonography over conventional breast sonography in detecting and localizing breast lesions by comparing the diagnostic accuracy of ductosonography and conventional breast sonography in detecting suspicious and unclear sonographic lesions.In Addition, reliability and time requirement of ductosonographic examination will be investigated. The second specific aim is to investigate the potential of tissue elasticity as a diagnostic marker in solid breast lesions (US-BI-RADS 3, 4 and 5) by elastosonography. The study design allows investigating the reproducibility of the method.

DETAILED DESCRIPTION:
The Research Project consists of mainly two parts that involve different methodological approaches: For the first part, different breast ultrasound techniques will be employed for the examination of an unselected population in a regular setting of a breast outpatient clinic. The second part includes measuring and characterizing tissue elasticity of breast lesions by elastosonography.

ELIGIBILITY:
Inclusion Criteria:all women , who agree with the two examinations of the breast: conventional method and ductosonography

Exclusion Criteria:

a women, who have only the conventional examination of sonography

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The recruitment of ductosonography will target all women attending the outpatient breast clinic of the department og gynecology and Obstretic, University of Basel, Switzerland.
Sampling Method: Non-Probability Sample
Enrollment: 236 (Actual)
Dates: Start 2011-08; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Improving Breast Cancer Diagnostic by Novel sonographicTechniques Study | 3 year and 6 months
  Comparing Time of Both Procedures of Conventional Sonography Versus Ductosonography Technique Elastosonography
Improving Breast Cancer Diagnostic by Novel sonographicTechniques Study | 3 year and 6 months
  Comparing the diagnostic accuracy of ductosonography and conventional breast sonography in the detection of breast lesions. Suspicious and unclear sonographic lesions (BI-RADS 3, 4, and 5) are clarified with a breast biopsy and malignancy confirmed by histology.

SECONDARY OUTCOMES:
Improving Breast Cancer Diagnostic by Novel sonographicTechniques Study | 3 year and 6 months
  Spatial precision will be evaluated by measuring the deviation in millimeters of sonographic detection sites from the site of the biopsy. Comparing the time requirement for ductosonography and traditional sonography in minutes

CONTACTS AND LOCATIONS:
Overall Officials: Rosanna Zanetti, PD Dr Med, Principal Investigator — Claraspital Basel
Locations (1):
- University Hospital of Basel, Basel, Canton of Basel-City, Switzerland

REFERENCES:
- [Derived] Brasier-Lutz P, Jaggi-Wickes C, Schaedelin S, Burian R, Schoenenberger CA, Zanetti-Dallenbach R. Agreement in breast lesion assessment and final BI-RADS classification between radial and meander-like breast ultrasound. BMC Med Imaging. 2021 Jun 22;21(1):104. doi: 10.1186/s12880-021-00632-1. PMID 34157997
- [Derived] Jaggi-Wickes C, Brasier-Lutz P, Schaedelin S, Burian R, Schoenenberger CA, Zanetti-Dallenbach R. Comparison of radial and meander-like breast ultrasound with respect to diagnostic accuracy and examination time. Arch Gynecol Obstet. 2020 Jun;301(6):1533-1541. doi: 10.1007/s00404-020-05554-x. Epub 2020 May 3. PMID 32363545